CLINICAL TRIAL: NCT00581958
Title: Radiation Biodosimetry in Patients Treated With Total Body Irradiation (TBI)
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Georgetown University (Other); National Institute of Standards and Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 07-158; NCT00899886 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Cancer
Keywords: total body irradiation; Cancer; Hematopoietic System
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine

GROUPS / COHORTS (1):
- Patients undergoing HSCT: Research subjects will have blood and/or urine sampled at three time points in the Department of Radiation Oncology. Participating patients will have at least a total two samples collected at each time point. The first sampling will occur before the first TBI treatment is given. The second sampling will occur before the second TBI treatment, usually 3 to 8 hours after the first treatment (in the case of multifraction TBI). If a patient is being treated with single fraction TBI, then the second sampling will occur approximately 3-8 hours after the first TBI treatment. The third and final sampling will occur at the next morning blood draw, prior to the fourth TBI treatment (in the case of multifraction TBI), 24 hours after the first TBI treatment.
  Interventions: Other: Blood Samples

INTERVENTIONS:
Other: Blood Samples — blood (approximately two 4 ml; equivalent to less than 2 tablespoon) and urine (a cup of urine) samples or testing a total of three times. Blood will be drawn and urine will be collected once before radiation treatment and twice after first radiation treatment.

SUMMARY:
The purpose of this study is to develop blood tests and urine tests that can tell doctors how much radiation a person has been exposed to. Doctors know how much radiation patients are exposed to in certain medical situations. An example of this would be radiation treatment for cancer. Radiation treatment machines are programmed to give exact doses of radiation.

DETAILED DESCRIPTION:
MSKCC patients undergoing TBI as part of a hematopoietic stem cell transplant (HSCT) will have blood drawn and urine collected for use in the validation and refinement of new methods for rapid high-throughput radiation biodosimetry. These blood and urine samples will be collected before, and at defined times after TBI. Blood sampling will occur in the same manner that it does during routine patient care during HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 4 years of age at Memorial Sloan-Kettering Cancer Center
* Must be undergoing hematopoietic stem cell transplantation (either autologous or allogenic) in conjunction with a conditioning regimen that includes TBI (single or multiple fraction)
* Functional central venous catheter

Exclusion Criteria:

* No subjects will be excluded from the proposed research study for demographic reasons. Treatment with growth factors, such as keratinocyte growth factor (KGF), will not be grounds for exclusion.
* Subjects who will receive radiation therapy within 5 days prior to TBI will be excluded.
* Subjects who will receive systemic antineoplastic chemotherapy within 7 days prior to TBI not have research bloods collected. Only urine will be collected from these patients.
* Based on current knowledge, we will not a priori exclude patients based on disease status (ie, patients in or out of remission will be included in this study), type of disease(ie, chromosomal breakage syndromes), or previous therapies (unless exclusion criteria is met).

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential research subjects will be identified by the primary Radiation Oncologist whom the patient is referred to by the Adult or Pediatric Bone Marrow Transplant Service.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
To develop, validate and refine high-throughput platforms for radiation biodosimetry using metabolomic assays. | 3 years
  The approach involves profiling blood and urinary metabolites that are specific for radiation exposure and dose.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Barker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Web Site — http://www.mskcc.org